CLINICAL TRIAL: NCT02559817
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Safety and Efficacy Study of a Range of Linaclotide Doses Administered Orally to Children, Ages 6 to 17 Years, A Multicenter, Randomized, Double-blind, Placebo-controlled Safety and Efficacy Study of a Range of Linaclotide Doses Administered Orally to Children Ages 7-17 Years, With Irritable Bowel Syndrome With Constipation (IBS-C) (ie, Fulfill Rome III Criteria for Child/Adolescent IBS and Fulfill Modified Rome III Criteria for Child/Adolescent Functional Constipation
Brief Title: A Safety and Efficacy Study of a Range of Linaclotide Doses Administered Orally to Children Ages 7-17 Years, With Irritable Bowel Syndrome With Constipation
Acronym: LIN-MD-63
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIN-MD-63
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Results first posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Irritable Bowel Syndrome With Constipation
Keywords: Irritable Bowel Syndrome with Constipation in children; Linzess
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Linaclotide Dose A (Experimental): Taken once daily each morning at least 30 minutes before breakfast, with the exception of the first Treatment Period dose which will be taken at the study center, after at least a 2-hour fast.
  Dose A: 18 micrograms liquid oral solution or solid oral capsule in children 7-11 years of age with weight 18 to <35 kg
  Dose A: 36 micrograms liquid oral solution or solid oral capsule in children 7-11 years of age with weight ≥ 35 kg
  Dose A: 36 micrograms solid oral capsule in children 12-17 years of age
  Interventions: Drug: Linaclotide Dose A
- Linaclotide Dose B (Experimental): Taken once daily each morning at least 30 minutes before breakfast, with the exception of the first Treatment Period dose which will be taken at the study center, after at least a 2-hour fast.
  Dose B: 36 micrograms liquid oral solution or solid oral capsule in children 7-11 years of age with weight 18 to <35 kg
  Dose B: 72 micrograms liquid oral solution or solid oral capsule in children 7-11 years of age with weight ≥ 35 kg
  Dose B: 72 micrograms solid oral capsule in children 12-17 years of age
  Interventions: Drug: Linaclotide Dose B
- Linaclotide Dose C (Experimental): Taken once daily each morning at least 30 minutes before breakfast, with the exception of the first Treatment Period dose which will be taken at the study center, after at least a 2-hour fast.
  Dose C: 72 micrograms liquid oral solution or solid oral capsule in children 7-11 years of age with weight 18 to <35 kg
  Dose C: 145 micrograms liquid oral solution or solid oral capsule in children 7-11 years of age with weight ≥ 35 kg
  Dose C: 145 micrograms solid oral capsule in children 12-17 years of age
  Interventions: Drug: Linaclotide Dose C
- Linaclotide Approved Adult Dose (Experimental): Taken once daily each morning at least 30 minutes before breakfast, with the exception of the first Treatment Period dose which will be taken at the study center, after at least a 2-hour fast.
  Approved Adult Dose: 290 micrograms solid oral capsule in children 12-17 years of age
  Interventions: Drug: Linaclotide Approved Adult Dose
- Matching Placebo (Placebo Comparator): Taken once daily each morning at least 30 minutes before breakfast, with the exception of the first Treatment Period dose which will be taken at the study center, after at least a 2-hour fast
  Placebo liquid oral solution or placebo solid oral capsule in children 7-11 years of age
  Placebo solid oral capsule in children 12-17 years of age
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Linaclotide Dose A
  Other Names: Linzess
  Arms: Linaclotide Dose A
Drug: Linaclotide Dose B
  Other Names: Linzess
  Arms: Linaclotide Dose B
Drug: Linaclotide Dose C
  Other Names: Linzess
  Arms: Linaclotide Dose C
Drug: Linaclotide Approved Adult Dose
  Other Names: Linzess
  Arms: Linaclotide Approved Adult Dose
Drug: Matching Placebo
  Other Names: Linzess
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of linaclotide for the treatment of Irritable Bowel syndrome with Constipation (IBS-C), in children age 7-17 years.

This study includes up to a 4-week Screening Period, and a 2 to 3-week Pretreatment Period. Patients age 7-11 will receive oral liquid or oral solid capsule and patients 12-17 will receive solid oral capsule formulation. Children ages 7-11 years meeting the entry criteria will be randomized to 1 of 3 doses of linaclotide or placebo for 4 weeks. Children ages 12-17 years meeting the entry criteria will be randomized to 1 of 4 doses of linaclotide or placebo for 4 weeks.

This 4-week study will assess the effects of linaclotide on bowel movement frequency, as well as other bowel symptoms of IBS-C.

ELIGIBILITY:
Inclusion Criteria:

* Patient weighs at least 18 kg (39.7 lbs)
* Patient meets Rome III criteria for child/adolescent IBS: at least once per week for at least 2 months before Screening Visit, the patient experienced abdominal discomfort (an uncomfortable sensation not described as pain) or pain associated with 2 or more of the following at least 25% of the time:
* a) Improvement with defecation
* b) Onset associated with a change in frequency of stool
* c) Onset associated with a change in form (appearance) of stool
* Patient meets modified Rome III criteria for child/adolescent Functional Constipation (FC): For at least 2 months before the Screening Visit, the patient has had 2 or fewer defecations (with each defecation occurring in the absence of any laxative, suppository, or enema use during the preceding 24 hours) in the toilet per week. In addition, at least once per week, patient meets 1 or more of the following:
* a) History of retentive posturing or excessive volitional stool retention
* b) History of painful or hard bowel movements (BMs)
* c) Presence of a large fecal mass in the rectum
* d) History of large diameter stools that may obstruct the toilet
* Patient is willing to discontinue any laxatives used before the Pretreatment Visit in favor of the protocol-permitted rescue medicine
* Patient has an average of fewer than 3 spontaneous BMs (SBMs) per week during the 14 days before the randomization day and up to the randomization. An SBM is defined as a BM that occurs in the absence of laxative, enema, or suppository use on the calendar day of the BM or the calendar day before the BM
* Patient or parent/guardian/LAR or caregiver is compliant with eDiary by completing both the morning and evening assessments for 10 out of the 14 days immediately preceding the Randomization Visit

Exclusion Criteria:

* Patient reports having more than 1 loose, mushy stool (eDiary-recorded stool consistency of 6 on the Pediatric Bristol Stool Form Scale [p-BSFS]) or any watery stool (eDiary-recorded stool consistency of 7 on the p-BSFS) with any SBM that occurred in the absence of laxative use on the calendar day of the BM or the calendar day before the BM during the 14 days before the randomization day and up to the randomization
* Select medical history or conditions that may be related to other causes of constipation or may interfere with safety and efficacy analyses
* Patient has required manual disimpaction anytime prior to randomization or disimpaction during in-patient hospitalization within one year prior to randomization
* Patient is unable to tolerate the placebo during rhe Screening Period

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Muslin, Study Chair — Forest Laboratories, LLC, an Allergan Affiliate
Locations (47):
- United States (45):
  - HealthStar Research, LLC, Hot Springs, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Advanced Research Center - Site 069, Anaheim, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - WCCT Global, LLC, Costa Mesa, California
  - ACTCA, Inc, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Center for Clinical Trials, LLC, Paramount, California
  - University of California at San Francisco, San Francisco, California
  - Advanced Medical Research Center, Miami, Florida
  - Children's Center for Digestive Health Care LLC, Atlanta, Georgia
  - Sleepcare Clinical Research Institute, Stockbridge, Georgia
  - Methodist Medical Center, Peoria, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Willis-Knighton Physician Network, Shreveport, Louisiana
  - Certified Research Consultants Virgo/Carter Pediatrics, Silver Spring, Maryland
  - GI Associates and Endoscopy Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Boys Town National Research Hospital, Boys Town, Nebraska
  - Midwest Children Health Research Institute, Lincoln, Nebraska
  - Goryeb Children's Hospital, Morristown, New Jersey
  - Columbia University Medical Center and Morgan Stanley Children's Hospital of New York, New York, New York
  - Asheboro Research Associates - Site 022, Asheboro, North Carolina
  - Capital Pediatrics and Adolescent Center PLLC, Raleigh, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ohio Pediatric Research Association, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Montgomery Medical Inc., Smithfield, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Coastal Pediatric Research, Charleston, South Carolina
  - Coastal Pediatrics Associates, Mt. Pleasant, South Carolina
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital/Baylor College Medicine, Houston, Texas
  - Houston Clinical Research Associates, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Tech Carilion School of Medicine Pediatric Gastroenterology, Roanoke, Virginia
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
  - Aurora Health Care, Aurora Medical Center in Summit, Summit, Wisconsin
- Canada (2):
  - Children's Hospital of Western Ontario, London, Ontario
  - Physician's Clinical Research Inc., Vaughan, Ontario

REFERENCES:
- [Derived] Di Lorenzo C, Nurko S, Hyams JS, Rodriguez-Araujo G, Shakhnovich V, Saps M, Simon M. Safety and efficacy of linaclotide in children aged 7-17 years with irritable bowel syndrome with constipation. J Pediatr Gastroenterol Nutr. 2024 Mar;78(3):539-547. doi: 10.1002/jpn3.12103. Epub 2023 Dec 28. PMID 38504394

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a screening period of 14 to 28 days, followed by a Pretreatment period of 14 to 21 days, prior to randomization of study participants.
Groups:
- Matching Placebo: Taken once daily each evening, at least 30 minutes before their evening meal, with the exception of the first Treatment Period dose which will be taken at the study center, after at least a 2-hour fast
  Placebo liquid oral solution or placebo solid oral capsule in children 7-11 years of age
  Placebo solid oral capsule in children 12-17 years of age
- Linaclotide Dose A: Taken once daily each evening, at least 30 minutes before their evening meal, with the exception of the first Treatment Period dose which will be taken at the study center, after at least a 2-hour fast.
  Dose A: 18 micrograms liquid oral solution or solid oral capsule in children 7-11 years of age with weight 18 to <35 kg
  Dose A: 36 micrograms liquid oral solution or solid oral capsule in children 7-11 years of age with weight ≥ 35 kg
  Dose A: 36 micrograms solid oral capsule in children 12-17 years of age
- Linaclotide Dose B: Taken once daily each evening, at least 30 minutes before their evening meal, with the exception of the first Treatment Period dose which will be taken at the study center, after at least a 2-hour fast.
  Dose B: 36 micrograms liquid oral solution or solid oral capsule in children 7-11 years of age with weight 18 to <35 kg
  Dose B: 72 micrograms liquid oral solution or solid oral capsule in children 7-11 years of age with weight ≥ 35 kg
  Dose B: 72 micrograms solid oral capsule in children 12-17 years of age
- Linaclotide Dose C: Taken once daily each evening, at least 30 minutes before their evening meal,, with the exception of the first Treatment Period dose which will be taken at the study center, after at least a 2-hour fast.
  Dose C: 72 micrograms liquid oral solution or solid oral capsule in children 7-11 years of age with weight 18 to <35 kg
  Dose C: 145 micrograms liquid oral solution or solid oral capsule in children 7-11 years of age with weight ≥ 35 kg
  Dose C: 145 micrograms solid oral capsule in children 12-17 years of age
- Linaclotide Approved Adult Dose: Taken once daily each evening, at least 30 minutes before their evening meal, with the exception of the first Treatment Period dose which will be taken at the study center, after at least a 2-hour fast.
  Approved Adult Dose: 290 micrograms solid oral capsule in children 12-17 years of age
Period: Treatment Period
Arm/Group | Matching Placebo | Linaclotide Dose A | Linaclotide Dose B | Linaclotide Dose C | Linaclotide Approved Adult Dose
Started | 19 | 29 | 21 | 24 | 8
Completed | 18 | 27 | 19 | 22 | 8
Not Completed | 1 | 2 | 2 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0
Not completed — Non-Compliance With Study Drug | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Period: Post-treatment Period
Arm/Group | Matching Placebo | Linaclotide Dose A | Linaclotide Dose B | Linaclotide Dose C | Linaclotide Approved Adult Dose
Started | 18 | 27 | 20 (1 participant who did not complete the first period, entered and completed the Post-treatment Period) | 22 | 8
Completed | 18 | 27 | 20 | 22 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 101 randomized participants took at least 1 dose of double-blind study treatment, which also comprises the Safety Population of 101 participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | Linaclotide Dose A | Linaclotide Dose B | Linaclotide Dose C | Linaclotide Approved Adult Dose | Total
Number analyzed (Participants) | 19 | 29 | 21 | 24 | 8 | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.9 (2.61) | 11.9 (2.95) | 12.7 (3.51) | 12.4 (3.26) | 13.5 (1.77) | 12.3 (3.00)
Age, Customized [Count of Participants; unit: Participants]
  Age: 7 years through 11 years | 8 | 13 | 9 | 11 | 0 | 41
  Age: 12 years through 17 years | 11 | 16 | 12 | 13 | 8 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 15 | 16 | 5 | 68
  Male | 6 | 10 | 6 | 8 | 3 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 17 | 15 | 16 | 6 | 66
  Black or African American | 7 | 10 | 6 | 7 | 1 | 31
  Multiple | 0 | 2 | 0 | 1 | 1 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 4 | 7 | 5 | 7 | 3 | 26
  Not Hispanic or Latino | 15 | 22 | 16 | 17 | 5 | 75
Weight [Mean (Standard Deviation); unit: kg] | 49.87 (14.387) | 55.22 (19.339) | 60.13 (22.670) | 56.80 (20.943) | 61.93 (17.586) | 56.14 (19.523)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.29 (3.266) | 23.56 (5.322) | 24.85 (6.304) | 24.57 (8.517) | 23.92 (5.955) | 23.67 (6.208)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 4-week Overall Spontaneous Bowel Movement (SBM) Frequency Rate (SBMs/Week) During the Treatment Period
Description: SBM was defined as a BM that occurred in the absence of laxative, suppository, or enema use on the calendar day of the BM or the calendar day before the BM. SBM rate was defined as SBMs/week during the 4-week Treatment period. Participants recorded the occurrence of BMs and use of rescue medication, morning and evening, daily in an eDiary since pretreatment period. The SBM frequency rate (SBMs/week) during the analysis period for each participant were calculated as [(total number of SBMs in the analysis period/number of days in the analysis period)*7]. Baseline value was based on values collected 14 days before randomization up to randomization. Change from Baseline was calculated as the SBM frequency rate during the 4-week treatment period - SBM frequency rate at baseline. A positive change from Baseline indicates improvement.
Time Frame: Baseline (14 days prior to randomization and up to randomization) to week 4
Population: ITT population, all participants who had at least 1 postbaseline entry on BM characteristic assessments that determined occurrences of SBMs (i.e. BM frequency and rescue medication use).
Measure: Mean (Standard Deviation); unit: Spontaneous Bowel Movements per Week
Arm/Group | Matching Placebo | Linaclotide Dose A | Linaclotide Dose B | Linaclotide Dose C | Linaclotide Approved Adult Dose
Number analyzed (Participants) | 19 | 29 | 21 | 23 | 8
Spontaneous Bowel Movements per Week | 1.447 (1.376) | 1.991 (2.349) | 2.298 (2.634) | 2.678 (2.774) | 3.222 (2.194)

2. Secondary Outcome: Change From Baseline in 4-week Abdominal Pain Daytime Symptoms Based on Evening Assessment of Abdominal Pain Symptoms
Description: The abdominal pain score was measured using 5-point scale. Participants answered the questions, How much did your tummy hurt as: 0=none, 1=a tiny bit, 2=a little, 3=some, and 4=a lot. The 4-week daytime abdominal pain was calculated as the average of nonmissing scores in evening eDiary during the Treatment Period with higher value indicating greater symptom severity. Baseline value was the average of non-missing values collected 14 days before randomization. Change from Baseline was calculated as the daytime abdominal pain score during the 4-week treatment period (i.e. average of non-missing daytime scores during 4-week treatment period) - daytime abdominal pain score at baseline. A negative change from Baseline indicates improvement.
Time Frame: Baseline (14 days prior to randomization) to week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Matching Placebo | Linaclotide Dose A | Linaclotide Dose B | Linaclotide Dose C | Linaclotide Approved Adult Dose
Number analyzed (Participants) | 19 | 29 | 21 | 23 | 8
Units on a Scale | -0.654 (0.789) | -0.709 (0.977) | -0.565 (0.861) | -0.648 (0.948) | -1.192 (1.032)

3. Secondary Outcome: Change From Baseline in 4-week Stool Consistency
Description: Participants used 7-point pediatric Bristol Stool Form (p-BSFS) scale to rate stool consistency for each BM in morning and evening eDiary where 1=small hard lumps or balls like pebbles,2=fat sausage shape but lumpy and hard,3=a sausage but with cracks on it,4=sausage or snake, smooth and soft,5=chicken nuggets, soft smooth blobs,6=oatmeal, fluffy mushy pieces,7=milkshake, watery. Scores in 4-week treatment period were calculated as mean of participants non-missing, SBM associated p-BSFS scores during 4-week treatment period. Baseline value was based on values collected 14 days before randomization up to randomization.
Time Frame: Baseline (14 days prior to randomization and up to randomization) to week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Matching Placebo | Linaclotide Dose A | Linaclotide Dose B | Linaclotide Dose C | Linaclotide Approved Adult Dose
Number analyzed (Participants) | 16 | 24 | 16 | 22 | 8
Units on a Scale | 0.653 (0.949) | 1.200 (1.068) | 1.502 (1.272) | 2.054 (1.349) | 1.345 (0.813)

4. Secondary Outcome: Change From Baseline in 4-week Severity of Straining
Description: Severity of straining was scored on 5-point scale for question-When you pooped, how hard did you push? The score ranges from 0= not hard at all,1= I pushed a tiny bit hard,2= I pushed a little hard,3= I pushed hard,4= I pushed very hard with higher scores indicating more severe straining. Participants recorded degree of straining for each BM in morning and evening eDiary. Scores during 4-week treatment period were calculated as mean of participant's non-missing, SBM associated straining scores during 4-week treatment period.
Time Frame: Baseline (14 days prior to randomization and up to randomization) to week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Matching Placebo | Linaclotide Dose A | Linaclotide Dose B | Linaclotide Dose C | Linaclotide Approved Adult Dose
Number analyzed (Participants) | 17 | 24 | 16 | 22 | 8
Units on a Scale | -0.576 (0.915) | -0.782 (1.187) | -0.859 (0.993) | -1.222 (0.972) | -1.236 (1.042)

5. Secondary Outcome: Change From Baseline in 4-week Abdominal Bloating Daytime Symptoms Based on Evening Assessment
Description: Participants recorded their assessment of abdominal bloating in the evening eDiary. Participants answered the question: How big and full did your tummy feel? on a scale, where: 0=none, 1=a tiny bit, 2=a little, 3=medium or 4=very, with a higher score indicating more severe bloating. Baseline value was the average of values collected 14 days before randomization. The 4-week daytime abdominal bloating symptoms were calculated as the average of non-missing scores reported in the evening eDiary during the treatment period. Change from Baseline was calculated as the 4-week daytime abdominal bloating score during the treatment period - daytime abdominal bloating score at baseline. A negative change from Baseline indicates improvement.
Time Frame: Baseline (14 days prior to randomization) to week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Matching Placebo | Linaclotide Dose A | Linaclotide Dose B | Linaclotide Dose C | Linaclotide Approved Adult Dose
Number analyzed (Participants) | 19 | 29 | 21 | 22 | 8
Units on a Scale | -0.438 (0.754) | -0.486 (0.974) | -0.515 (0.992) | -0.440 (0.823) | -0.595 (1.284)

6. Secondary Outcome: Change From Baseline in 4-week Overall Complete Spontaneous Bowel Movement (CSBM) Frequency Rate (CSBMs Per Week)
Description: SBM was defined as a BM that occurred in the absence of laxative, suppository, or enema use on the calendar day of the BM or the calendar day before the BM. A CSBM was an SBM that was associated with a sense of complete evacuation. Participants recorded their assessment of the sensation of incomplete evacuation for each BM in the morning and evening eDiary. The 4-week overall CSBM frequency rate was calculated as [total number of CSBMs in the analysis period/number of days in the analysis period]*7). Baseline value was based on values collected 14 days before randomization and up to randomization. Change from Baseline was calculated as the CSBM frequency rate during the 4-week treatment period - CSBM frequency rate at baseline. A positive change from Baseline indicates improvement.
Time Frame: Baseline (14 days prior to randomization and up to randomization) to week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CSBMs per Week
Arm/Group | Matching Placebo | Linaclotide Dose A | Linaclotide Dose B | Linaclotide Dose C | Linaclotide Approved Adult Dose
Number analyzed (Participants) | 19 | 29 | 21 | 23 | 8
CSBMs per Week | 0.825 (1.211) | 0.644 (1.029) | 1.167 (1.822) | 1.721 (2.292) | 2.358 (2.199)

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment period (4 weeks), up to Day 30 after the last dose, for serious adverse events (SAEs) and all-cause mortality. From the first dose, up to Day 1 after the last dose, for other adverse events.
Arm/Group | Matching Placebo | Linaclotide Dose A | Linaclotide Dose B | Linaclotide Dose C | Linaclotide Approved Adult Dose
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/29 | 0/21 | 0/24 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/29 | 0/21 | 0/24 | 0/8
Other Adverse Events (participants affected / at risk) | 3/19 | 6/29 | 5/21 | 3/24 | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Matching Placebo (N=19) | Linaclotide Dose A (N=29) | Linaclotide Dose B (N=21) | Linaclotide Dose C (N=24) | Linaclotide Approved Adult Dose (N=8)
Anaphylactic Reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Matching Placebo (N=19) | Linaclotide Dose A (N=29) | Linaclotide Dose B (N=21) | Linaclotide Dose C (N=24) | Linaclotide Approved Adult Dose (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 3 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to slow participant enrollment, further screening was terminated. This decision was not due to any safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study are the property of the Sponsor. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and the Sponsor and will follow the Sponsor's standard operating procedures on publications.

DOCUMENTS (2):
  • Study Protocol (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT02559817/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT02559817/SAP_001.pdf